CLINICAL TRIAL: NCT07245641
Title: Targeted Accelerated TMS for Post-Traumatic Stress Disorder
Acronym: TAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Mass General Home Base Program (Unknown)
Responsible Party: Principal Investigator, Joseph J. Taylor, MD, PhD, Clinical Director of TMS, Center for Brain Circuit Therapeutics, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P002359
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
Keywords: Accelerated Transcranial Magnetic Stimulation; Post traumatic stress disorder; PTSD; TMS; Neuromodulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel-group double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to receive either 1) active aTMS at their individualized target or 2) sham aTMS at their individualized target in a 2:1 randomization. One research assistant (RA) is the only individual unblinded in this study. The unblinded RA will have no other interactions with participants. RAs delivering treatment with stimulate participants with sham or active aTMS, with randomization assigned by the unblinded RA. Blind will be broken at 1-month follow-up visit for all participants, physicians, and treating technicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active aiTBS (Active Comparator): Participants in this group will receive active aiTBS with neuronavigation to a treatment target identified with individualized resting state functional connectivity.
  Interventions: Procedure: Transcranial Magnetic Stimulation
- Sham aiTBS (Sham Comparator): Participants in this group will receive sham aiTBS with neuronavigation to a treatment target identified with individualized resting state functional connectivity. Participants in the sham group who continue to present with moderate PTSD symptoms (greater than or equal to 33 cutoff on PCL-5) at the post-treatment month 1 visit will be offered the opportunity to opt in and receive another course of active aTMS.
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a focal, non-invasive form of brain stimulation that has FDA clearance for depression. In this study, a form of TMS called accelerated intermittent theta burst stimulation (aiTBS) will be administered under the supervision of a physician with TMS expertise.
  Other Names: TMS; Accelerated intermittent theta burst stimulation; aiTBS

SUMMARY:
Post-traumatic stress disorder (PTSD) is a highly prevalent and debilitating condition among veterans and active-duty military personnel, with rates as high as 30% in certain combat-exposed populations. Conventional treatments such as prolonged exposure therapy and pharmacotherapy have limited efficacy and high dropout rates, highlighting the need for novel, rapidly effective interventions.

Transcranial magnetic stimulation (TMS) has been well established for treatment-resistant depression (TRD). Traditional TMS, which involves 6 to 7 weeks of daily, weekday scalp-targeted treatment, shows open-label response and remission rates of 58.1% and 30%, respectively. However, such protocols may be impractical for military personnel with limited medical leave. A new form of accelerated TMS (aTMS) that involves 10 imaging-guided treatments per day for 5 consecutive days has demonstrated substantial antidepressant benefits within days and response rates of 69% at 1-month follow-up. This protocol has not been tested for PTSD, in part because there was no causally informed brain circuit target. In this study, the investigators will test aTMS for PTSD using a novel PTSD circuit that the investigators have derived.

DETAILED DESCRIPTION:
In a recent study in Nature Neuroscience, the investigators analyzed three independent datasets to derive a brain circuit causally linked to PTSD in military veterans. Investigators found that brain lesions that reduce the probability of developing PTSD (n=193) were connected to the same brain circuit based on the functional connectivity profiles of individual patients with PTSD using fMRI (n=180). Finally, investigators demonstrated that scalp-targeted TMS to our circuit rapidly improved PTSD symptoms (n=20).

Separately, the investigators partnered with a private clinic to administer open-label, circuit-targeted aTMS to patients with PTSD (n=8). Investigators found that the treatment was safe and tolerable. Response and remission rates were 75% and 63%, respectively. Of note, these response and remission rates assess outcomes up to 4 weeks after the treatment ends. This approach captures individual variability in response trajectory and aligns with our own data from aTMS treatment of TRD.

The strength of these findings has inspired us to launch a pilot randomized controlled aTMS trial in which the investigators prospectively target our PTSD circuit using each patient's neuroimaging data in combination with the accelerated TMS treatment protocol.

ELIGIBILITY:
Inclusion Criteria

* Age 18-65
* DSM-5 diagnosis of PTSD per PTSD Checklist for DSM-5 (CAPS-5)
* At least moderate symptoms of PTSD per PCL-5 (≥21)
* English proficiency sufficient to understand risks/benefits
* No new medications or medication increases before, during, or after aTMS
* Primary clinician (e.g. psychiatrist, therapist, psychologist, APRN, PA, etc.) responsible for psychiatric care before, during, and after the trial
* Agreement to lifestyle considerations:
* Abstain from becoming pregnant from screening to one-month after treatment (the MRI visit)
* Continue usual intake patterns of caffeine- or xanthine-containing products (e.g. coffee, tea, soft drinks, chocolate) throughout treatment
* No changes to routine intake of alcohol, tobacco, and recreational drugs if patients are using them at baseline for at least 24 hours before the start of each MRI and TMS session

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist with Criterion A for DSM-5 (PCL-5) | Before treatment to 1-month post treatment
  20 item PTSD scale, scored 0-80. Higher scores indicate worse symptoms. Investigators will use a repeated measures mixed model to examine the effect of treatment on PCL-5 scores over time as well as a group x time interaction not controlling for depression.
  Hypothesis: There will be a significant difference in PCL-5 score magnitude of change one month after treatment relative to baseline in the participants receiving active treatment vs. sham

SECONDARY OUTCOMES:
PTSD Checklist with Criterion A for DSM-5 (PCL-5) | Before treatment to 1-month post treatment
  20 item PTSD scale, scored 0-80. Higher scores indicate worse symptoms. Investigators will determine between-group effect size based on the change in PCL-5 score one month after treatment.
  Hypothesis: Relative to sham aTMS, active aTMS will show a moderate-to-large effect size.

OTHER OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAP-5) | Before treatment and 1 month after treatment
  30-item clinical interview designed to assess PTSD based on DSM-5 criteria. Total scores from 0-80, with higher numbers indicating greater PTSD symptom severity.
Clinically Useful Anxiety Outcome Scale (CUXOS) | Before treatment and daily for 5 treatment days
  20-item, self-report questionnaire that measures the severity of psychic and somatic anxiety symptoms. Scores range from 0-80, which higher scores indicating higher symptoms of anxiety.
Beck Depression Inventory (BDI) | Before treatment, 1 week post treatment, and 1 month post treatment
  Depression severity rating scales (0-63, higher numbers indicate higher severity)
Beck Anxiety Inventory (BAI) | Before treatment, 1 week post treatment, and 1 month post treatment
  Anxiety severity rating scale (0-63, higher numbers indicate higher severity)
Young Mania Rating Scale (YMRS) | Before treatment, daily for 5 treatment days, and 1 month post treatment
  11 item scale evaluating mania. Scored 0-60. Higher score indicates worse outcome/higher mania
Patient Global Impressions (PGI) | Before and 1 month after treatment
  A single question assessing a patient's perception of their health or condition. Scores range from 1-7, one being the participant believes they are not at all ill, seven being an extremely ill individual.
Clinical Global Impression Scale (CGI) | Before and 1 month after treatment
  Clinician-rated tool to assess the global severity of a patient's illness. 7-point scale from 1 (very much improved) to 7 (very much worse).
Adult Temperament Questionnaire | Before treatment and 1 month after treatment
  77-item self-report questionnaire assessing individuals temperament and personality. Scores range from 0-539, with scores in subsections of the questionnaire indicating various affects and temperaments.
World Health Organization Disability Assessment Schedule II (WHODAS 2.0) | Before treatment and 1 month after treatment
  36-item functional assessment (each question rated 1-5) Minimum: 36 Maximum: 180 Can also be scored by percentiles Higher score indicates more disability
World Health Organization Quality of Life (WHOQOL-BREF) | Before treatment and 1 month after treatment
  26-item questionnaire assessing an individual's perception of their quality of life (scores range from 0 to 100, where higher scores represent a better quality of life).
Visual Analog Scale (Mood) | Before treatment and daily for 5 treatment days
  A single question asking participants to rate their current mood on a scale of 1-100 (higher scores indicate positive mood)
Adult Attention Deficit/Hyperactivity Disorder Self-Report Scale (AARS) | Before treatment and 1 month after treatment
  ADHD rating scale (each question rated 1-5, higher scores indicate symptoms highly consistent with ADHD)
Illness Intrusiveness Rating Scale (IIRS) | Before treatment and 1 month after treatment
  3 item scale measuring how illness affects function. Scored 13-91, higher score indicates higher illness intrusiveness severity
McLean Screening Instrument for Borderline Personality Disorder (MS-BPD) | Before treatment and 1 month after treatment
  10-item questionnaire used to screen for BPD (scores range from 0 to 10; higher scores are associated with higher levels of/more severe BPD symptoms).
Perceived Stress Scale (PSS) | Before treatment and 1 month after treatment
  Stress assessment scored 0-40, higher scores indicate higher stress
Social Readjustment Rating Scale (SRRS) | Before and 1 month after treatment
  A tool used to assess the potential stress associated with different life events (scores range from 0 to 430, with higher scores indicating higher levels of stress).
Pittsburgh sleep quality index (PSQI) | Before and 1 month after treatment
  Self-report questionnaire to assess sleep quality, scored from 0 to 21. Higher scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carpenter LL, Janicak PG, Aaronson ST, Boyadjis T, Brock DG, Cook IA, Dunner DL, Lanocha K, Solvason HB, Demitrack MA. Transcranial magnetic stimulation (TMS) for major depression: a multisite, naturalistic, observational study of acute treatment outcomes in clinical practice. Depress Anxiety. 2012 Jul;29(7):587-96. doi: 10.1002/da.21969. Epub 2012 Jun 11. PMID 22689344
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Siddiqi SH, Philip NS, Palm ST, Carreon DM, Arulpragasam AR, Barredo J, Bouchard H, Ferguson MA, Grafman JH, Morey RA, Fox MD. A potential target for noninvasive neuromodulation of PTSD symptoms derived from focal brain lesions in veterans. Nat Neurosci. 2024 Nov;27(11):2231-2239. doi: 10.1038/s41593-024-01772-7. Epub 2024 Sep 24. PMID 39317797
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062